CLINICAL TRIAL: NCT02356263
Title: Adaptation and Validation of Recent Life Changes Questionnaire (RLCQ) to Measure Stress Among Adult Population of Karachi, Pakistan.
Brief Title: Adaptation and Validation of Recent Life Changes Questionnaire for Measuring Stress Among Adults in Karachi, Pakistan
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Associate Professor Neurology,Director Stroke Fellowship Program, Aga Khan University
Other Study IDs: 3235-CHS-ERC-14
Record Dates: First submitted 2015-01-28; First posted 2015-02-05 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Life Change Events
Keywords: stressful events; psychological stress; life experiences
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Stressors impair optimum function of an individual physiologically and psychologically. Overcoming stress is possible when one knows which aspects of life are the most troublesome to manage for individuals. There are certain tools available in Pakistan that can measures stress in selected populations but there are no validated tools that may quantify stress which results from events occurring in different aspects of life.

Recent Life Changes Questionnaire (RLCQ) is a tool that measures stress of individuals through life changing events. It has five categories; work, home and family, health, personal and social and financial. The objective of the study is to adapt RLCQ and validate it so that it may measure stress among people living in Karachi, Pakistan.

DETAILED DESCRIPTION:
In order to make RLCQ a tool to measure stress within Pakistani context, we would want to adapt RLCQ and then validate it. The study design is a validation study where the construct of recent life changing events will be validated by comparing it with a gold standard to assess the extent of accuracy of measurement by exploring the agreement between them. The mode of data collection is cross-sectional by administering the adapted RLCQ and the gold standard simultaneously. Since stress is a subjective phenomenon and serves as a root cause for many neurodegenerative diseases and mental disorders, a tool for screening mental illnesses is selected against which we could compare the adapted RLCQ for validation. The Mini international neuropsychiatric Interviews (MINI) is a structured diagnostic interview developed and validated by Sheehan in 1997, Florida. It is based on the DSM IV criteria and ICD-10. The design of this study incorporates content and criterion validity as we have a pre-existing 'gold standard' which is widely accepted and is in current practice of mental health screening in Pakistan.

The study will be conducted in six phases. Phase I includes conducting qualitative interviews to explore the phenomenon. In Phase II, adaptation of RLCQ will be done and review of the adapted tool will be done with the help of subject experts. Phase III will verify the face validity of the tool by translations and back translations. In Phase IV, pre-testing of the tool will be done whereas in phase V, we will administer the tool in the community along with conducting MINI interviews. Phase VI tests the reliability of the tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* Those who would stay in the study site for at least one month
* Those who provide a written informed consent

Exclusion Criteria:

* Those who do not understand Urdu
* Those who have cognitive or hearing difficulties
* People with known psychiatric conditions and are under treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the study includes all adults aged 18 years or above living in Karachi, Pakistan. The source population is that of all adults aged 18 years or above living in Gulshan-e-Iqbal town Karachi from where we will draw our sample population comprising of those adults 18 years or more who fulfil the eligibility criteria and consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity, as measured by Positive and Negative Predictive Value, Kappa Statistics | 11 months
  sensitivity and specificity of the RLCQ will be compared against gold standard MINI

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Derived] Artani A, Kamal AK, Azam SI, Artani M, Bhamani SS, Saif M, Khan FA, Alam N. Validation of the Recent Life Changes Questionnaire (RLCQ) for stress measurement among adults residing in urban communities in Pakistan. BMC Psychol. 2019 Oct 21;7(1):66. doi: 10.1186/s40359-019-0341-9. PMID 31639054
- [Derived] Artani A, Bhamani SS, Azam I, AbdulSultan M, Khoja A, Kamal AK. Adaptation of the Recent Life Changes Questionnaire (RLCQ) to measure stressful life events in adults residing in an urban megapolis in Pakistan. BMC Psychiatry. 2017 May 5;17(1):169. doi: 10.1186/s12888-017-1315-1. PMID 28476102